CLINICAL TRIAL: NCT03601689
Title: Predictive Factors of Disease-free Survival After Complete Pathological Response to Neoadjuvant Radiotherapy in Rectal Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Moroccan Society of Surgery (Other)
Responsible Party: Sponsor
Other Study IDs: CompleteResponse
Record Dates: First submitted 2018-07-14; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Rectal Neoplasms
Keywords: Low rectal cancer; Neoadjuvant treatment; Complete pathological response; ypT0N0; disease free survival; Predictive factors
MeSH Terms: conditions — Rectal Neoplasms; Pathologic Complete Response | interventions — Proctectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: rectal resection — total mesorectal excision

SUMMARY:
Many data suggest that patients with low rectal adenocarcinoma who achieved ypT0N0 status have improved survival and disease-free survival (DFS) compared to all other stages however only few data are available regarding the specific prognosis factors of this subgroup. This retrospective multicentric study aimed to predict the prognosis of patients with complete pathological response after neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria

* patients with a histologically proven low rectal adenocarcinoma,
* no previous or synchronous colorectal disease,
* UICC stage I-III patients who underwent neoadjuvant chemoradiotherapy or chemotherapy,
* followed by total mesorectal excision (TME), and
* a complete pathological response defined as ypT0N0

Exclusion Criteria:

- all patients with metastatic tumors or missing data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who underwent neoadjuvant treatment followed by total mesorectal excision for rectal adenocarcinoma in 8 centers
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Local recurrence rate | From date of surgery until the date of first documented local progression assessed up to 100 months
  A postoperative local recurrence was defined by biopsy-proven or radiographic evidence of local recurrent disease.
Distant recurrence rate | From date of surgery until the date of first documented distant progression assessed up to 100 months
  A postoperative distant recurrence was defined by biopsy-proven or radiographic evidence of distant recurrent disease.

SECONDARY OUTCOMES:
Predictive factors of disease free survival | From date of surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Disease free survival was defined as the period between the day of surgery and the date of recurrence or the last date of follow-up

CONTACTS AND LOCATIONS:
Locations (8):
- Batna anticancer center, Algiers, Algeria
- Morocco (7):
  - Mohammed V University Medical School, Surgery Department, Military Hospital, Rabat, Please Enter the State Or Province
  - Mohammed V University Medical School, Surgical Department "A", Ibn Sina Hospital, Rabat, Please Enter the State Or Province
  - Mohammed V University Medical School, Surgical Department "C", Ibn Sina Hospital,, Rabat, Please Enter the State Or Province
  - National Institut of Oncology, Surgical oncology department, Rabat, Please Enter the State Or Province
  - Sidi Mohammed Ben Abdellah University Medical School, Surgery Department,, Fes
  - Mohammed Ist University Medical School, Surgical Oncology, Hospital el Farabi, Oujda
  - Private surgical oncology center, Salé

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Souadka A, Majbar MA, Benkabbou A, Serji B, Souiki T, Bouchentouf SM, Abid M, El Khannousi B, El Harroudi T, El Malki HO, Raiss M, Ifrine L, Mazaz K, Zentar A, Mohsine R, Souadka A, Belkouchi A, Ahallat M, Hrora A; Moroccan Society of Surgery. Predictive factors of disease-free survival after complete pathological response to neoadjuvant radiotherapy for rectal adenocarcinoma: retrospective case series. BMC Cancer. 2019 Oct 28;19(1):1008. doi: 10.1186/s12885-019-6239-3. PMID 31660903